CLINICAL TRIAL: NCT06188143
Title: The Efficacy of Combination of Ibuprofen and Paracetamol for Pain Control in Diagnostic Hysteroscopy
Brief Title: Study of Pain Control in Diagnostic Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PMK-019
Record Dates: First submitted 2023-12-10; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No medication before hysteroscopic procedure
- Ibuprofen-Paracetamol (Experimental): Ibuprofen 40mg and Paracetamol 500mg per oral, single dose each, before hysteroscopic procedure 30minutes
  Interventions: Combination Product: Ibuprofen-Paracetamol

INTERVENTIONS:
Combination Product: Ibuprofen-Paracetamol — Ibuprofen 40mg and Paracetamol 500mg per oral, single dose each, in study group 30minutes before hysteroscopic procedure
  Arms: Ibuprofen-Paracetamol

SUMMARY:
The goal of this clinical trial study is to learn about how to decrease the pain during the diagnostic hysteroscopy. The main question it aims to answer is "Do the Paracetamol and Ibuprofen taken before the procedure can lower the pain during the diagnostic hysteroscopy".

DETAILED DESCRIPTION:
After the participants those are indicated for diagnostic hysteroscopy and eligible for the study undergo informed consent, then they were divided to two groups for control group those get no medication and study group those get Paracetamol 500mg and Ibuprofen40mg per oral before the hysteroscopy, and both group needs to evaluate the pain score in VAS before, during hysteroscopy and after hysteroscopy for 30 minutes to compare the pain level in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with indication and informed to undergo diagnostic hysteroscopy over or equal the age of 20 years old

Exclusion Criteria:

* Women with contraindication for undergoing diagnostic hysteroscopy includes women with pregnancy, uterine infection, diagnosed with cervical cancer or endometrium cancer and women who is undergoing with active vaginal bleeding
* Women with history of allergy to Paracetamol or Ibuprofen medicine
* Women with currently or pre-existing medical conditions that contraindicate the use of ibuprofen includes kidney disease, heart disease, cirrhosis, gastritis or individuals with a history of peptic ulcer or gastrointestinal bleeding
* Women with currently taking anticoagulant or antiplatelet medications
* Women with history of psychiatric disorders

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 58 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
The pain score comparing between study and control group | During and 30minutes after the hysteroscopic procedure
  Comparing the pain score in visual analogue scale of 1(minimum) to 10scores(maximum) which is less to more painful respectively(higher score means more painful and worse outcome)

SECONDARY OUTCOMES:
The associated factors effecting the pain of the procedure | During and 30minutes after the hysteroscopic procedure
  Comparing the pain score in visual analogue scale of 1(minimum) to 10scores (maximum) which is less to more painful respectively(higher score means more painful and worse outcome)between the participants with the possible associated factor effecting the pain of the procedure those are history of undergo vaginal delivery, history of undergo the hysteroscopy procedure and post menopause in both control group(no medication) and study group(Paracetamol and Ibuprofen)

CONTACTS AND LOCATIONS:
Locations (1):
- Phramongkutklao College of Medicine and Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No